CLINICAL TRIAL: NCT06176131
Title: Implementering af Cardiostafet tværsektoriel Samarbejdsmodel Med Telemedicin for Udsatte Patienter Med Hjertesvigt Som Ikke Kan Deltage i Hjerterehabilitering
Brief Title: The Cardio-share Telemedicine Cross-sector Collaboration Model for Managing Vulnerable Patients With Heart Failure
Acronym: ADHFQUAL-BFH
Status: Recruiting | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Helena DOMINGUEZ, Consultant, Associate Professor, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: WorkZone-23072092
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure，Congestive; Atrial Fibrillation
Keywords: heart failure; atrial fibrillation; acute decompensated heart failure; heart failure with reduced ejection fraction; heart failure with preserved ejection fraction; telemedicine; health inequity; cross-sector health management
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cardio-share: Patients with successful cardio-share model fulfill at least one of the following:
  1. A plan for follow-up after discharge established, based on communication with Primary Care (home-care and/or General Practice) before discharge
  2. The patient has accessed MinSP-Ass. and received information on heart failure
  3. The patient has sent vital measurements and symptoms through MinSP-Ass. to the hospital cardiologist
  Interventions: Other: Telemedicine-based cross-sector collaboration for patient management
- Others: All others who fulfill the inclusion criteria but none of the three elements have been successful are the comparative group "Others"

INTERVENTIONS:
Other: Telemedicine-based cross-sector collaboration for patient management — Telemedicine support from the hospital-based cardiology heart-failure team is provided on demand defined by the needs from Primary Care and from the patient rather than plain guideline-based targets
  Groups: cardio-share

SUMMARY:
The goal of this observational study is to explore the potential of implementing a telemedicine-based cross-sector collaboration model to manage patients with frequent admissions with decompensated heart failure. The main question(s) it aims to answer are:

* Characterization of conditions that make these patients vulnerable
* Description of key-elements that makes possible to manage the patients with the cardio-share model

Participants are:

* Patients - will be helped to use the available telemedicine tools
* General Practitioners - will be offered teleconferences with cardiologists (chat and video) on demand
* Community health workers (caregivers at the patient home or in elderly home) - will be guided to assist the patients to use the available telemedicine tools Researchers will compare readmission rates (primary outcome) and quality of life of patients where the cardio-share management model is successfully implemented one year before and after the implementation.

DETAILED DESCRIPTION:
Consecutive patients admitted from 01.01.2024 to one single site (University Hospital Bispebjerg and Frederiksberg) with acute decompensated heart failure or with atrial fibrillation treated with loop-diuretics will be included in the project if they had one emergency admission with decompensated heart condition within the prior 3 months or two or more within the prior 6 months.

During their hospital admission patients will be helped to use the currently available telemedicine tools, which is "Min Sundhedsdplatformen Assistent" (MinSP-Ass.), which is the Danish version of the Care Companion-extension of MyChart application by EPIC, which is the platform used in East Denmark. Help is provided by the nurses in the ward, with assistance by medicine students working on a pay-per-hour basis.

The cardio-share model briefly If it is planned or the patient already is receiving home-care assistance (either at home or at an elderly home), the health-care workers will be contacted to ensure that they can assist the patient to use MinSP-Ass.

Likewise, the general practice where the patient belongs to, will be contacted to offer teleconsultation support by the hospital-based cardiologist. This support is primarily by written messages, and by teleconferences on demand (from Primary Care) before patient discharge, in both cases using MedCom standards, which is the current cross-sector communication platform in Denmark.

Through MinSP-Ass. patients can receive educational material and can report vital measurements and symptoms.

The responsibility of the management of the patient relays in the hospital cardiologist who initiates the cardio-share management. A script for a seamless switching of this responsibility between the cardiologist team and Primary Care will be developed and described throughout the project. This will include solving data-sharing across sectors since there are no current solutions easy to use for this purpose.

Data collection The electronic medical record will be explored retrospectively to record data at three time-points: After discharge (Baseline), three and six months after admission.

At baseline there will be recorded: i) demography data, ii) selected vital measurements and laboratory data and iii) heart medicines.

At month three there will be recorded whether there has been at least one readmission and the date of the first readmission and if the patient has had visits in the cardiology ambulatory. At month six there will be recorded whether there have been one or more readmissions and the date of the first readmission if it occurred after month 3.

Demography data will be collected according to the following conditions that may render the patient vulnerable:

* Speaking Danish language
* Cognitive challenges described in the medical record
* Need for help from health community workers or relatives for their daily life
* Psychiatric disease (ongoing follow-up)
* Substance abuse (alcohol or drugs)

At baseline and at month 6 there will be recorded:

* Selected vital measurements, which include blood pressure, heart rate and weight
* Laboratory data, which include hemoglobin, creatinine and pro-Brain Natriuretic Peptide (pro-BNP)
* Prescription and use of heart medicines

ELIGIBILITY:
Inclusion Criteria:

Patients admitted with acute decompensated heart failure AND:

* with previous admission with decompensated heart failure in the three-month period prior to the current admission or
* who have two or more admissions in the 6 months prior to the current admission.

Exclusion Criteria:

* Patients who

  * have refused to share their data for health-quality projects
  * have already ongoing telemedicine management for heart failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the University Hospital of Bispebjerg and Frederiksberg and for whom this is their reference hospital for general heart conditions.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Days out-of-hospital | six months
  Number of days out of hospital from date of discharge for the index event until the next re-admission with acute decompensated heart failure

SECONDARY OUTCOMES:
Number of readmissions | six months
  number of emergency readmissions after discharge from the index readmission, where there have been signs of decompensated heart failure
Quality of care - Medicines | six months
  Proportion of guideline-based target medicines for heart failure that patients actually use (based on purchased medicine prescriptions). This includes angiotensin converter enzyme inhibitors(ACEi)/angiotensin receptor blockers (ARB), Betablockers, Mineralocorticoids, Angiotensin Receptor Neprilysin inhibitors (ARNi), Selective Sodium Glucose Co-Transporter-2 inhibitors (SGLT2i), Hydralazine and Nitrates.
Symptom-based quality of care | six months
  Progression of heart failure specific patient-reported outcome measures. These include weekly to monthly collected: • Out-of-breath in daily activities • Night orthopnea • Dizziness • Feeling body fluid retention (leg swelling, increased abdominal pressure, increased intake of diuretics • Tiredness • Feeling of general worsening

OTHER OUTCOMES:
Palliative care | six months
  Number of subjects with established palliative care

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Wisborg, MD,PhD,DrM, Study Director — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Cardiology department Y, Bispebjerg-Frederiksberg Hospital, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided